CLINICAL TRIAL: NCT04402801
Title: Impact on Patient Outcomes of Clinic Transition From Face to Face Encounters to Telemedicine in the Cystic Fibrosis (CF) Adult Population at UVA
Brief Title: Patient Outcomes of Clinic Transition From Face to Face Encounter to Telemedicine in Cystic Fibrosis
Status: Completed | Type: Observational
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Dana Albon, MD, Assistant Professor, University of Virginia
Other Study IDs: 22327
Record Dates: First submitted 2020-05-20; First posted 2020-05-27 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Standard of Care Telemedicine Cohort: This cohort will have telemedicine visits in lieu of in-person clinic visits
- Standard of Care In-Person Cohort

SUMMARY:
Adult patients with Cystic Fibrosis who are seen at the specialty CF clinic at University of Virginia will be given an option to utilize telemedicine instead of in-person visits for standard clinic visits. Health information from standard of care visits including FEV1, exacerbations, leading to oral or intravenous antibiotics, laboratory results, hospitalization records, and responses to health questionnaires will be recorded for research purposes. Data collected for the research study will be compared to baseline and previous years to determine if there are any deleterious effects for those who transition to telemedicine clinic visits.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18-year-old and older) with CF seen in the UVA adult CF clinic who agree to participate in the study.

Exclusion Criteria:

* Patients who cannot consent to the research study. In addition, prisoners will not be included.

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult CF patients 18 yo and older.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
FEV1 stability | 12 months
  A change of 10% or more in FEV1 percent predicted will be considered significant; FEV1 pre and pos covid telemedicine implementation will be compared

SECONDARY OUTCOMES:
Exacerbation rate | 12 months
  Exacerbation rate pre and pos covid telemedicine implementation will be compared

CONTACTS AND LOCATIONS:
Overall Officials: Dana Albon, MD, Principal Investigator — University of Virginia Health System
Locations (1):
- University of Virginia Health System, Charlottesville, Virginia, United States

REFERENCES:
- [Result] Somerville LAL, List RP, Compton MH, Bruschwein HM, Jennings D, Jones MK, Murray RK, Starheim ER, Webb KM, Gettle LS, Albon DP. Real-World Outcomes in Cystic Fibrosis Telemedicine Clinical Care in a Time of a Global Pandemic. Chest. 2022 May;161(5):1167-1179. doi: 10.1016/j.chest.2021.11.035. Epub 2021 Dec 10. PMID 34896356
- [Derived] Bruschwein HM, Soper M, Jennings D, Somerville L, List R, Compton MH, Turner R, Albon D. Mental health screening of patients with cystic fibrosis through telehealth during COVID-19: Evaluation of feasibility and process adoption. Fam Syst Health. 2022 Sep;40(3):397-402. doi: 10.1037/fsh0000698. Epub 2022 May 23. PMID 35604723